CLINICAL TRIAL: NCT03611790
Title: The Vesalio Neva VS for the Treatment of Symptomatic Cerebral Vasospasm Following Aneurysmal Subarachnoid Hemorrhage (aSAH) (The VITAL Study)
Brief Title: Vesalio NeVa VS for Symptomatic Cerebral Vasospasm Following aSAH (The VITAL Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-002 / D
Record Dates: First submitted 2018-07-18; First posted 2018-08-02 (Actual); Results first posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): NeVa VS
  Interventions: Device: NeVa VS

INTERVENTIONS:
Device: NeVa VS — mechanical dilatation

SUMMARY:
The objective of the study is to assess the safety and probable benefit of the Neva VS device in patients presenting with symptomatic cerebral vasospasm despite maximal medical management following aSAH.

DETAILED DESCRIPTION:
This is a prospective, open label, single-arm study. Up to 30 eligible subjects at up to 15 sites will participate in the study. Subjects will be followed up for 30 days post-intervention.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Subarachnoid hemorrhage secondary to ruptured aneurysm.
* Ruptured aneurysm secured with surgical clipping or endovascular intervention.
* Digital subtraction angiography (DSA) or CT angiography at the time of aSAH clinical presentation or aSAH intervention with well-visualized intra-cerebral vessels is available for review.
* Vasospasm in one or more of the following: the internal carotid artery (ICA), basilar, middle cerebral artery (MCA), anterior cerebral artery (ACA), or posterior cerebral artery (PCA) territory on transcranial Doppler (TCD), and/or CT angiography, and/or clinical signs of symptomatic vasospasm (change in level of consciousness, focal neurological deficit) confirmed by > 50% narrowing in these territories on DSA.
* Vasospasm despite maximized medical management defined as oral Nimodipine (unless contraindicated), systemic hypertension with SBP greater than 130 mmHg and euvolemia.
* Target vessel pre-vasospasm diameter ≥ 2 mm and ≤ 4.0 mm.
* Subject or legal representative is able and willing to give informed consent.

Exclusion Criteria

* The presence of an unsecured ruptured aneurysm. Note unsecured unruptured aneurysms remote to the site of treated aSAH are not an exclusionary.
* Symptoms attributable to other causes (e.g., hydrocephalus, metabolic, infection).
* Hunt and Hess Grade of 5
* Large infarct on CT scan defined as ASPECTS 0-5.
* Intracranial hemorrhage not caused by aneurysm rupture.
* History of bleeding disorders.
* Baseline platelets < 30,000.
* International normalized ratio (INR) > 1.7.
* Any known contraindications to mechanical dilation of vasospastic vessels including but not limited to:
* Excessive vessel tortuosity that prevents the placement of the device
* Evidence of rapidly improving neurological signs of stroke
* Large territory completed cerebral infarction, edema with mass effect and intra-parenchymal hemorrhage in vascular territory to be treated, or
* any other vascular anatomic variants or anomalies
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor (e.g. Aricept).
* History of severe allergy to contrast medium.
* Known allergy to NeVa materials (nitinol, stainless steel).
* Suspected or confirmed septic embolus, or bacterial endocarditis.
* Septic shock or central nervous system (CNS) infection confirmed via cerebrospinal fluid (CSF) sampling.
* Known current or recent use of illicit drugs or alcohol abuse.
* Females who are pregnant or breastfeeding.
* Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure is performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - RIA Neurovascular Clinic, Englewood, Colorado
  - Baptist Health System, Jacksonville, Florida
  - Wellstar Health System, Marietta, Georgia
  - University of Buffalo, Buffalo, New York
  - North Shore University Hospital - Northwell, Manhasset, New York
  - Mount Sinai Health System, New York, New York
  - SUNY Stony Brook University, Stony Brook, New York
  - Fort Sanders Regional Med Center, Knoxville, Tennessee
  - TTUHSC El Paso, El Paso, Texas
  - Houston Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 51.8 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: defined as 50% or greater vessel caliber on DSA compared to baseline, as determined by the core laboratory
Time Frame: within 30 minutes of completion of procedure
Population: The VITAL study data were analyzed using descriptive statistics due to the small sample size (N=30).
Measure: Count of Units; unit: Vessels Treated
Units Other Than Participants: Vessels Treated
Groups:
- Single Arm - NeVa VS Intervention: NeVa VS Intervention
Arm/Group | Single Arm - NeVa VS Intervention
Number analyzed (Participants) | 30
Number analyzed (Vessels Treated) | 74
Vessels Treated | 64

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Single Arm - NeVa VS Intervention
All-Cause Mortality (participants affected / at risk) | 7/30
Serious Adverse Events (participants affected / at risk) | 17/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - NeVa VS Intervention (N=30)
Intraprocedural thrombotic event (Vascular disorders) | 2 (2)
Cerebral infarct (Vascular disorders) | 1 (1)
Cerebral infarct secondary to vasospasm (Vascular disorders) | 1 (1)
Pseudoaneurysm of the contralateral femoral artery (Vascular disorders) | 1 (1)
Ruptured vessel due to balloon angioplasty (Vascular disorders) | 1 (1)
Worsening cardiomyopathy (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Cerebral infarct secondary to vasospasm (Vascular disorders) | 3 (3)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Cerebral hemorrhage secondary to right ventriculostomy catheter removal (Vascular disorders) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pseudoaneurysm of the brachial artery (Vascular disorders) | 1 (1)
Recurrent SAH (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Worsening ascites (Gastrointestinal disorders) | 1 (1)
Worsening hydrocephalus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - NeVa VS Intervention (N=30)
Intraprocedural thrombotic event (Vascular disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 8 (8)
Anemia post-24 hours (Blood and lymphatic system disorders) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 5 (6)
Cerebral salt wasting syndrome (Nervous system disorders) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Cerebral infarct secondary to vasospasm (Vascular disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data resulting from this study is the proprietary information of the Sponsor. None of the data resulting from this study will be allowed to be presented or published in any form, by the investigator or any other person, without the prior written approval of the Sponsor.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03611790/Prot_SAP_ICF_000.pdf